CLINICAL TRIAL: NCT00731211
Title: A Phase II Trial of Pazopanib in Patients With Metastatic Renal Cell Carcinoma Previously Treated With Sunitinib or Bevacizumab
Brief Title: Pazopanib in Previously Treated Patients With Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GU 56
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Results first posted 2015-05-20 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; Metastatic; Pazopanib; Previously-treated
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pazopanib (Experimental): 800 mg of pazopanib orally each day continuously
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — 800 mg of pazopanib orally each day continuously
  Other Names: Votrient

SUMMARY:
This is a Phase II, non-randomized, open-label, single-arm study in patients with metastatic renal cell carcinoma who have received one prior targeted therapy with either sunitinib or bevacizumab. The planned enrollment for this study is 60 patients.

DETAILED DESCRIPTION:
All eligible patients will receive 800 mg of pazopanib orally each day continuously. Patients will be re-evaluated for treatment response after 8 weeks of daily oral pazopanib therapy. Response to therapy will be assigned using RECIST criteria (Section 6.0) Patients who have objective response or stable disease will continue treatment with evaluations every 8 weeks, until the time of tumor progression or intolerable treatment-related side effects.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have histologically documented metastatic or unresectable locally recurrent clear cell renal carcinoma. In patients with mixed histologies, any percentage of clear cell histology is acceptable.
2. Patients must have had only one previous targeted agent therapy with either sunitinib or bevacizumab. Patients must have progressed either during or within 3 months of discontinuing treatment with one of these agents. Patients who stopped either sunitinib or bevacizumab because of unacceptable toxicity are also eligible.
3. Patients may have received one previous regimen containing traditional immunotherapy (interferon, interleukin-2), chemotherapy, or combination chemoimmunotherapy for metastatic disease.
4. Previous nephrectomy is required unless clinically contraindicated (e.g. extensive liver or bone metastases; primary tumor <5cm).
5. An ECOG performance status of 0 or 1.
6. At least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques, or as >10 mm with spiral computerized tomography (CT) scan according to the Response Evaluation Criteria in Solid Tumors (RECIST).
7. Absolute neutrophil count (ANC) >1500; platelets >75,000 (within 7 days prior to study treatment).
8. Adequate liver function as measured by serum bilirubin <1.5 mg/dL and AST/ALT <2.5 times upper limit of normal (ULN) (or <5 x ULN in patients with documented liver metastases).
9. Serum creatinine <2.0 mg/dL.
10. Patients must be able to understand the nature of this study and give written informed consent.

Exclusion Criteria:

1. Previous treatment with more than one targeted agent, or more than one previous traditional regimen (e.g., chemotherapy, immunotherapy, chemoimmunotherapy).
2. Previous treatment with sorafenib, temsirolimus, everolimus or other investigational targeted agents.
3. Inability to swallow and retain oral medication.
4. History of other malignancy. Patients who have been disease-free for 5 years, or patients with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
5. Concurrent disease or condition that would make the patient inappropriate for study participation including: (1) any unresolved or unstable serious toxicity from prior administration of another drug, or (2) any serious medical disorder that would interfere with the patient's safety, obtaining informed consent, or compliance with the study.
6. History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously treated parenchymal CNS metastases, are asymptomatic, and have had no requirement for steroids or anticonvulsants for >2 months prior to study enrollment. Routine screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required only if clinically indicated, or if the patient has a history of CNS metastases.
7. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel.
8. Active peptic ulcer disease, inflammatory bowel disease, or other gastrointestinal condition increasing the risk of perforation.
9. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 4 weeks prior to beginning therapy.
10. Presence of uncontrolled infection.
11. Concurrent cancer therapy (e.g., chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, hormonal therapy, or tumor embolization).
12. Concurrent treatment with an investigational agent or participation in another clinical trial.
13. Use of an investigational anti-cancer drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of pazopanib.
14. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib.
15. Has taken or is taking prohibited medications.
16. Corrected QT interval (QTc) prolongation defined as QTc interval >470 msec.
17. History of any one of the following cardiac conditions within the past 6 months:

    * Cardiac angioplasty or stenting
    * Myocardial infarction
    * Unstable angina
    * History of cerebrovascular accident within the past 6 months
    * Poorly controlled hypertension (systolic blood pressure [SBP] of >140 mmHg, or diastolic blood pressure [DBP] of >90 mmHg).

    Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. The blood pressure (BP) must be re- assessed on two occasions that are separated by a minimum of 24 hours. The mean SBP-DBP values from both BP assessments must be <140/90 mmHg in order for a patient to be eligible for the study.
18. Presence of any non-healing wound, fracture, or ulcer, or the presence of symptomatic peripheral vascular disease.
19. Evidence of bleeding diathesis or coagulopathy.
20. Major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks prior to beginning therapy, or anticipation of the need for a major surgical procedure during the course of the study. Minor surgical procedures such as fine needle aspiration or core biopsy within 1 week prior to beginning therapy are also excluded.
21. Pregnant or lactating female. All patients of childbearing potential must agree to use adequate contraception for 2 weeks prior to beginning pazopanib, during the entire study, and for 60 days after pazopanib is discontinued.
22. Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
23. History of untreated deep venous thrombosis (DVT) within the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-09; Primary Completion 2011-05 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Hainsworth, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (17):
- United States (17):
  - San Francisco Oncology Associates, San Francisco, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Watson Clinic Center for Cancer Care and Research, Lakeland, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Gulfcoast Oncology Associates, St. Petersburg, Florida
  - Medical Oncology Associates of Augusta, Augusta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Baptist Hospital East, Louisville, Kentucky
  - Central Maine Medical Center, Lewiston, Maine
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - St. Louis Cancer Care, Chesterfield, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Oncology Hematology Care, Cincinnati, Ohio
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Virginia Cancer Institute, Richmond, Virginia

REFERENCES:
- [Result] Hainsworth JD, Rubin MS, Arrowsmith ER, Khatcheressian J, Crane EJ, Franco LA. Pazopanib as second-line treatment after sunitinib or bevacizumab in patients with advanced renal cell carcinoma: a Sarah Cannon Oncology Research Consortium Phase II Trial. Clin Genitourin Cancer. 2013 Sep;11(3):270-5. doi: 10.1016/j.clgc.2013.04.006. Epub 2013 May 9. PMID 23665131

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pazopanib
Started | 55 (2 patients ineligible (papillary histologic type-1 pt. Previous treatment with everolimus alone-1 pt)
Completed | 55
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All eligible patients
Arm/Group | Pazopanib
Number analyzed (Participants) | 55
Age, Continuous [Median (Full Range); unit: years] | 60 [41 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 42
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Proportion of patients with complete and partial response (CR and PR). CR defined as disappearance of target lesions; PR defined as at least a 30% decrease in the sum of the longest diamater of target lesions.
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Pazopanib
Number analyzed (Participants) | 55
percentage of patients | 27 [17 to 40]

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is measured from Day 1 of study drug administration to disease progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or death on study. Progression is defined in RECIST v1.1 as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: every 8 weeks until progressive disease, expected average of 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pazopanib
Number analyzed (Participants) | 55
months | 7.5 [5.4 to 9.4]

ADVERSE EVENTS:
Arm/Group | Pazopanib
Serious Adverse Events (participants affected / at risk) | 10/55
Other Adverse Events (participants affected / at risk) | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib (N=55)
Nervous system disorders - Other, speech impairment (Nervous system disorders) | 1 — event
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Headache (Nervous system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Psychiatric disorders - Other, change in mental status (Psychiatric disorders) | 1
Hypertension (Vascular disorders) | 1
Gastrointestinal disorders - Other, hemorrhage (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Hematoma (Vascular disorders) | 1
General disorders and administration site conditions - Other, failure to thrive (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib (N=55)
Alkaline phosphatase increased (Investigations) | 5
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 5
Alanine aminotransferase increased (Investigations) | 14
Anorexia (Metabolism and nutrition disorders) | 19
Aspartate aminotransferase increased (Investigations) | 13
Blood bilirubin increased (Investigations) | 6
Blurred vision (Eye disorders) | 7
Skin and subcutaneous tissue disorders - Other, burning skin (Skin and subcutaneous tissue disorders) | 3
Confusion (Psychiatric disorders) | 4
Constipation (Gastrointestinal disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Creatinine increased (Investigations) | 13
Dehydration (Metabolism and nutrition disorders) | 8
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 14
Diarrhea (Gastrointestinal disorders) | 34
Dizziness (Nervous system disorders) | 8
Dry skin (Skin and subcutaneous tissue disorders) | 4
Dysphagia (Gastrointestinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18
Edema face (General disorders) | 7
Edema limbs (General disorders) | 17
Fatigue (General disorders) | 45
Fever (General disorders) | 6
Flatulence (Gastrointestinal disorders) | 4
Skin and subcutaneous tissue disorders - Other, hair changes (Skin and subcutaneous tissue disorders) | 3
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 5
Anemia (Blood and lymphatic system disorders) | 23
Gastrointestinal disorders - Other, hemorrhage (Gastrointestinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Renal and urinary disorders - Other, urinary hemorrhage (Renal and urinary disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 13
Hyperkalemia (Metabolism and nutrition disorders) | 7
Hypertension (Vascular disorders) | 22
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 6
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 7
Lip infection (Infections and infestations) | 3
Infections and infestations - Other, oral infection (Infections and infestations) | 4
Upper respiratory infection (Infections and infestations) | 6
Insomnia (Psychiatric disorders) | 8
White blood cell decreased (Investigations) | 6
Memory impairment (Nervous system disorders) | 4
Depression (Psychiatric disorders) | 6
Mucositis (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 33
Peripheral sensory neuropathy (Nervous system disorders) | 15
Abdominal pain (Gastrointestinal disorders) | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 19
Bone pain (Musculoskeletal and connective tissue disorders) | 8
Non-cardiac chest pain (General disorders) | 4
Toothache (Gastrointestinal disorders) | 3
Headache (Nervous system disorders) | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18
Myalgia (Musculoskeletal and connective tissue disorders) | 11
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Pain (General disorders) | 5
Oral pain (Gastrointestinal disorders) | 5
Platelet count decreased (Investigations) | 14
Proteinuria (Renal and urinary disorders) | 25
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 18
Gastroesophageal reflux disease (Gastrointestinal disorders) | 10
Skin and subcutaneous tissue disorders - Other, skin changes (Skin and subcutaneous tissue disorders) | 11
Nervous system disorders - Other, speech impairment (Nervous system disorders) | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5
Dysgeusia (Nervous system disorders) | 17
Eye disorders - Other, vision changes (Eye disorders) | 3
Vomiting (Gastrointestinal disorders) | 13
Watering eyes (Eye disorders) | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 10
Weight loss (Investigations) | 12
Wound complication (Injury, poisoning and procedural complications) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites